CLINICAL TRIAL: NCT04106011
Title: Cognitive Changes Associated With Initiation of Gabapentin Treatment in Adults With Chronic Pain
Brief Title: Cognitive Changes With Gabapentin Treatment
Status: Terminated | Type: Observational
Why Stopped: PI request - low enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jessica Justmann, Instructor, Washington University School of Medicine
Other Study IDs: 201908050
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Neuralgia Peripheral; Pain
MeSH Terms: conditions — Pain | interventions — Gabapentin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Neuropathic Pain
  Interventions: Drug: Gabapentin; Diagnostic Test: BTACT; Diagnostic Test: BPI; Diagnostic Test: HADS; Diagnostic Test: SLP9; Diagnostic Test: NPSI

INTERVENTIONS:
Drug: Gabapentin — Titration of gabapentin will be standardized as 300mg QHS and increased by 300mg every 3 days until taking 1200mg TID or maximum tolerable dose. Subjects will undergo cognitive evaluation prior to initiation of the medication, at 1 week (when titrated to approximately 900mg/day), 3 weeks (when titrated to approximately 2100mg/day), and at 6 weeks (when titrated to 3600mg/day or maximum tolerable dose).
Diagnostic Test: BTACT — Cognition measure: Brief Test of Adult Cognition by Telephone
Diagnostic Test: BPI — Pain severity and interference at baseline using the Brief Pain Inventory
Diagnostic Test: HADS — Assessment of depression and anxiety with the Hospital Anxiety and Depression Scale
Diagnostic Test: SLP9 — Assessment of Sleep
Diagnostic Test: NPSI — Assessment of neuropathic components

SUMMARY:
This is a single-cohort, prospective, observational study evaluating the effects of gabapentin on cognition. The goal of the study is to determine whether there is a measurable change in cognitive function from baseline in patients who are prescribed gabapentin for the treatment of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85
2. Diagnosis of neuropathic pain
3. Patient report of average daily pain intensity in the last week >3 on 0-10 Numerical Rating Scale (NRS).
4. Able and willing to sign an IRB-approved written informed consent

Exclusion Criteria:

1. Current pregabalin treatment
2. Patient has started taking a new pain medication, or has changed their pain medication dose, in the past 4 weeks.
3. Treatment with opioids exceeding 60mg MME.
4. Severe cognitive impairment that is documented in medical chart.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic pain, who are prescribed gabapentin per standard of care
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Change in the Brief Test of Adult Cognition by Telephone (BTACT) | up to 6 weeks after treatment initiation
  Measure of cognitive functioning that assesses multiple dimensions central for effective functioning across adulthood: episodic memory, working memory, reasoning, verbal fluency, and executive functioning.
  Scoring:
  Word List Recall - Immediate & Delayed Total number unique is total number of correct responses (range 0-15)
  Backward Digit Span Score is highest number of digits reached (range 0, 2-8)
  Category Fluency Total number unique is total number of correct responses
  Red/Green Accuracy Normal baseline score is total number correct in normal baseline condition (range 0-20) Number Series Total number of items correct (range 0-5)
  Backward Counting Last number reached Total number of errors Total number of digits produced is calculated as: 100 - (number reached + number errors)

SECONDARY OUTCOMES:
Change in pain severity - BPI | up to 6 weeks after treatment initiation
  Medical questionnaire used to measure pain, developed by the Pain Research Group of the WHO Collaborating Center for Symptom Evaluation in Cancer Care 0-10 pain severity scale, 0=no pain, 10=pain as bad as you can imagine (scoring-a mean severity score) 0-10 pain relief scale, 0%=no relief, 100%=complete relief (only one question) 0-10 pain interference scale, 0=does not interfere, 10=completely interferes (scoring-mean of 7 items)
Change in Depression and Anxiety - HADS | up to 6 weeks after treatment initiation
  Measure of anxiety and depression in a general population of patients. Popular for clinical practice and research.
  Score- 8-10 mild, 11-14 moderate, 15-21 severe (separate scores for anxiety and depression)
Change in Sleep Problems - SLP9 | up to 6 weeks after treatment initiation
  Questionnaire to evaluate problems with sleep. Scale: 1=all of the time, 2=most of the time, 3=a good bit of the time, 4=some of the time, 5=a little of the time, 6=none of the time
  Final scores range from 0-100, with higher scores indicating more sleep problems. To score the SPI II, you must first transform the responses of each item into a new score. For item 1, responses of 1, 2, 3, 4, and 5 are scored as 0, 25, 50, 75, and 100, respectively. For items 3 and 9, ratings of 1 through 6 are scored as 0, 20, 40, 60, 80, and 100, respectively. All of the other items are reverse-scored (lower ratings indicate more sleep difficulties) and so ratings of 1 through 6 for these items are scored as 100, 80, 60, 40, 20, and 0, respectively. The final SPI II score is an average of the item scores responded to.
Change in Neuropathic Pain - NPSI | up to 6 weeks after treatment initiation
  Questionnaire to evaluate the different symptoms of neuropathic pain. 0-10 scale, 0=no sensation, 10=greatest sensation intensity

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justmann, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center/Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Berger A, Sadosky A, Dukes E, Edelsberg J, Oster G. Clinical characteristics and patterns of healthcare utilization in patients with painful neuropathic disorders in UK general practice: a retrospective cohort study. BMC Neurol. 2012 Mar 6;12:8. doi: 10.1186/1471-2377-12-8. PMID 22394606
- [Background] Finnerup NB, Attal N. Tapentadol prolonged release in the treatment of neuropathic pain related to diabetic polyneuropathy--authors' reply. Lancet Neurol. 2015 Jul;14(7):685-6. doi: 10.1016/S1474-4422(15)00060-5. No abstract available. PMID 26067119
- [Background] Fleet JL, Dixon SN, Kuwornu PJ, Dev VK, Montero-Odasso M, Burneo J, Garg AX. Gabapentin dose and the 30-day risk of altered mental status in older adults: A retrospective population-based study. PLoS One. 2018 Mar 14;13(3):e0193134. doi: 10.1371/journal.pone.0193134. eCollection 2018. PMID 29538407